CLINICAL TRIAL: NCT06166862
Title: Effect of Action Observation and Motor Imagery Therapy on Balance, Functional Status and Quality of Life in Stroke, Randomized Controlled Trial
Brief Title: Action Observation and Motor Imagery Therapy in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yurdagül Bahran Muştu, M.D., Principal investigator, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-2023/02
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation and motor imagery therapy for rehabilitation (Experimental): Action observation and motor imagery therapy for rehabilitation in stroke patients in addition to conventional rehabilitation programs.
  Interventions: Other: Action observation and motor imagery therapy for rehabilitation
- Sham action observation and motor imagery therapy for rehabilitation (Sham Comparator): Sham comparator for action observation and motor imagery therapy for rehabilitation in stroke patients in addition to conventional rehabilitation programs.
  Interventions: Other: Sham action observation and motor imagery therapy for rehabilitation

INTERVENTIONS:
Other: Action observation and motor imagery therapy for rehabilitation — Action observation; Patients will watch some exercises accompanied by music from a previously prepared video for 10 minutes. Exercises include 8-10 repetitions of abduction-adduction, horizontal abduction-adduction, flexion-extension and supination-pronation movements for the upper extremity, and stepping, forward-backward stepping, side stepping and ankle dorsiflexion movements for the lower extremity.
  Motor imagery training; Patients will be asked to visualize the actions they watched in their minds for 10 minutes.
  Then the patients will watch the video again and will be asked to perform the exercises while watching.
  Arms: Action observation and motor imagery therapy for rehabilitation
Other: Sham action observation and motor imagery therapy for rehabilitation — Sham action observation; Patients will watch a video consisting of static nature photographs for 10 minutes with the same music.
  Sham motor imaginary; Patients will think about the video they watched for 10 minutes.
  Then, they will watch another video in which the exercises are performed only once, and they will be asked to do the exercises. They will be given enough time to do 8-10 repetitions.
  Arms: Sham action observation and motor imagery therapy for rehabilitation

SUMMARY:
In recent years, motor imagery (MI) and action observation (AO) therapy strategies have been used in rehabilitation programs to increase motor learning in stroke. Visuomotor training strategies such as AO and MI therapy rely on the activity of the mirror neuron system to facilitate motor re-learning. Mirror neurons are activated during the performance of goal-directed actions, also when observing the same action and visualizing the action in the mind.

This clinical trial aims to test whether the application of AO and MI treatment in stroke in addition to conventional rehabilitation programs has an additional effect on motor recovery, activities of daily living, and quality of life.

DETAILED DESCRIPTION:
Stroke is one of the most common neurological disorders that causes chronic disability in adulthood. Stroke-related neurological dysfunction causes impairment in motor and sensory skills and limitation in the ability to perform daily living activities, resulting in decreased independence of patients. This process causes significant impairment in the quality of life of stroke patients.

In recent years, motor imagery (MI) and action observation (AO) therapy strategies have been used in rehabilitation programs to increase motor learning in stroke. Visuomotor training strategies such as AO and MI therapy rely on the activity of the mirror neuron system to facilitate motor re-learning. Mirror neurons are activated during the performance of goal-directed actions, also when observing the same action and visualizing the action in the mind.

This clinical trial aims to test whether the application of AO and MI treatment in stroke in addition to conventional rehabilitation programs has an additional effect on motor recovery, activities of daily living, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a stroke in the last year
* Functional Ambulation Classification score 2-5

Exclusion Criteria:

* Patients who have had repeated strokes
* Patients with neglect
* Patients with cognitive dysfunction (those who cannot follow simple verbal instructions)
* Patients with severe hearing problems
* Patients with severe vision problems
* Patients with additional musculoskeletal system pathology that will affect physical performance (such as amputation, severe joint mobility limitation, peripheral nerve damage)
* Patients with uncontrolled hypertension and diabetes mellitus
* Patients with a history of symptomatic lung disease (such as asthma, chronic obstructive pulmonary disease, emphysema)
* Patients with a history of symptomatic cardiac disease (such as coronary artery disease, arrhythmia, heart failure)
* Patients with peripheral artery disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The difference in the scores of the Fugl-Meyer Assessment between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Fugl-Meyer Assessment between pre- and post-rehabilitation assessments.
  The Fugl-Meyer Assessment is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The motor domain is used in this study, which includes items assessing movement, coordination, and reflex action of the upper and lower extremities. Motor score ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity.
The difference in the scores of the Brunnstrom stages between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Brunnstron stages between pre- and post-rehabilitation assessments.
  Brunnstrom staging assesses the motor recovery process of the hemiplegic patient in 6 stages (Stages 1 to 6). Upper extremity, lower extremity, and hand are evaluated separately. Higher stages indicate better motor function.

SECONDARY OUTCOMES:
The difference in the scores of the Barthel Index between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Barthel Index between pre- and post-rehabilitation assessments.
  The Barthel Index measures the functional independence of a person in mobility and activities of daily living. The index yields a total score out of 100 (0 to 100). The higher the score, the greater the degree of functional independence.
The difference in the scores of the Stroke-Specific Quality of Life Scale between pre- and post-rehabilitation | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Stroke-Specific Quality of Life Scale between pre- and post-rehabilitation assessments.
  Stroke Specific Quality of Life Scale assesses health-related quality of life specific to stroke survivors. It consists of a total of 49 items and the total score ranges from 49-245. Higher scores indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagul Bahran Mustu, MD., Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Karaman, Turkey (Türkiye)